CLINICAL TRIAL: NCT05457244
Title: A Prospective, Single-Center Investigation of the Safety and Performance of the da Vinci SP® Surgical System in Colorectal Procedures
Brief Title: Safety and Performance of the da Vinci SP® Surgical System in Colorectal Procedures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGMH-SP2021-4
Record Dates: First submitted 2022-06-22; First posted 2022-07-13 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Cancer; Robotic Surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Participant arm (Experimental)
  Interventions: Device: single-port robotic surgery

INTERVENTIONS:
Device: single-port robotic surgery — Colorectal surgery using the da Vinci SP System will be performed via the umbilicus, McBurney's site or the reverse McBurney's site depending on the sites of lesion. All of these patients will undergo a standard minimally invasive resection in the same fashion as would be carried out with multiport laparoscopic or robotic surgery.
  Other Names: da Vinci SP System

SUMMARY:
The study is a prospective, single-center, single-arm unblinded clinical investigation. The aim of this study is to evaluate the performance and safety of da Vinci SP system. This study will entail a collection of demographics, preoperative, perioperative and postoperative outcomes of the patients into a database to follow this report on the outcomes, and notably answer questions to demonstrate the performance and safety of this surgical option.

All patients being considered for minimally invasive colorectal surgery will be evaluated for participation in the above study. All of these patients will undergo a standard minimally invasive resection in the same fashion as would be carried out with multiport laparoscopic or robotic surgery

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Pathological confirm of colon or rectal cancer
* Clinical stage I-III
* Patient is a candidate for minimally invasive right hemicolectomy or anterior resection.
* ASA ≤3
* Performance status: ECOG 0-1

Exclusion Criteria:

* Emergency surgery
* Patient has metastatic disease
* Patient has a bleeding or clotting disorder
* Uncontrolled illness, including active infection, symptomatic heart failure, unstable angina or cardiac arrhythmias, or psychiatric illness that would limit compliance with study requirements
* Previous laparotomy history
* Patient unable to provide informed consent
* Patient is pregnant
* BMI 35.0 or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate (%) | immediately after the surgery
  Calculating the percentage of cases successfully performed using the da Vinci SP system via the SP access port with or without an additional 12mm assistant port. Conversion to laparoscopy or laparotomy will be considered as failure.

SECONDARY OUTCOMES:
Perioperative Parameters:Incision length | immediately after the surgery
  Incision length
Perioperative Parameters:Time of surgery | immediately after the surgery
  Time of surgery
Perioperative Parameters:Total operative time | immediately after the surgery
  Total operative time
Perioperative Parameters:Robotic console time | immediately after the surgery
  Robotic console time
Perioperative Parameters: Blood transfusions | immediately after the surgery
  Blood transfusion amount
Perioperative Parameters: Estimated blood loss | immediately after the surgery
  Estimated blood loss
Perioperative Parameters: Intra-operative Complications | immediately after the surgery
  Satava System
Perioperative Parameters: Urine output | immediately after the surgery
  Urine output
Perioperative Parameters: Type of anastomosis | immediately after the surgery
  How the anastomosis was performed and method of construction
Postoperative Parameters:pain requirements | Within 30days after the surgery
  type, frequency, total amount of narcotics used postoperatively per day
Postoperative Parameters:Pain score | Within 30days after the surgery
  NRS
Postoperative Parameters:Time to tolerate diets | Within 30days after the surgery
  time to tolerate clear liquids and solid food
Postoperative Parameters:Time to flatus | Within 30days after the surgery
  Time to flatus
Postoperative Parameters:Time to discharge | Within 30days after the surgery
  Time to discharge
Postoperative Parameters:Complications | Within 30days after the surgery
  Clavien-Dindo Classification
Postoperative Parameters:Readmission and reoperation rate | Within 30days after the surgery
  Readmission and reoperation rate

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chang Lu, MD, Principal Investigator — Kaohsiung Chang Gung Memorial
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marks J, Ng S, Mak T. Robotic transanal surgery (RTAS) with utilization of a next-generation single-port system: a cadaveric feasibility study. Tech Coloproctol. 2017 Jul;21(7):541-545. doi: 10.1007/s10151-017-1655-3. Epub 2017 Jul 14. PMID 28707106
- [Result] Kneist W, Stein H, Rheinwald M. Da Vinci Single-Port robot-assisted transanal mesorectal excision: a promising preclinical experience. Surg Endosc. 2020 Jul;34(7):3232-3235. doi: 10.1007/s00464-020-07444-4. Epub 2020 May 11. PMID 32394173
- [Result] Lin YM, Chen HH, Chen YJ, Chen PH, Lu CC. Single-incision laparoscopic colectomy using self-made glove port for benign colon diseases. J Laparoendosc Adv Surg Tech A. 2013 Nov;23(11):932-7. doi: 10.1089/lap.2013.0383. Epub 2013 Oct 11. PMID 24117036
- [Result] Lu CC, Lin SE, Chung KC, Rau KM. Comparison of clinical outcome of single-incision laparoscopic surgery using a simplified access system with conventional laparoscopic surgery for malignant colorectal disease. Colorectal Dis. 2012 Apr;14(4):e171-6. doi: 10.1111/j.1463-1318.2011.02825.x. PMID 21914101
- [Result] Lai WH, Lin YM, Lee KC, Chen HH, Chen YJ, Lu CC. The application of McBurney's single-incision laparoscopic colectomy alleviates the response of patients to postoperative wound pain. J Laparoendosc Adv Surg Tech A. 2014 Sep;24(9):606-11. doi: 10.1089/lap.2014.0167. Epub 2014 Jul 31. PMID 25079975
- [Result] Kim SJ, Choi BJ, Lee SC. Comparative analysis of outcomes after multiport and single-port laparoscopic colectomy in emergency situations: Is single-port laparoscopic colectomy safe and feasible? Asian J Surg. 2018 Jan;41(1):20-29. doi: 10.1016/j.asjsur.2016.07.008. Epub 2016 Aug 31. PMID 27592126